CLINICAL TRIAL: NCT01887626
Title: An Open-label, Randomised, 3-period, 3-treatment, Crossover, Single-centre, Single-dose, Bioavailability Study With Alternative Methods of Administration of Crushed Ticagrelor Tablets, 90 mg, Compared to Whole Ticagrelor Tablets, 90 mg, in Healthy Volunteer
Brief Title: Study to Investigate if the Uptake of Ticagrelor Into the Body Differs Depending on Method of Administration.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: D5130C00076
Record Dates: First submitted 2013-06-25; First posted 2013-06-27 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Bioavailability Heathy Volunteers
Keywords: Phase 1, pharmacokinetic, safety, Ticagrelor
MeSH Terms: interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Ticagrelor 90 mg as a whole tablet
  Interventions: Drug: Ticagrelor 90 mg whole tablet
- B (Experimental): Ticagrelor 90 mg tablet crushed and suspended in water
  Interventions: Drug: Ticagrelor 90 mg tablet crushed
- C (Experimental): Dispersed ticagrelor 90 mg tablet suspended in water and administered through a nasogastric tube into the the stomach
  Interventions: Drug: Dispersed ticagrelor 90 mg tablet suspended in water - nasogastric tube

INTERVENTIONS:
Drug: Ticagrelor 90 mg whole tablet — Ticagrelor 90 mg whole tablet administered as a single oral dose
  Arms: A
Drug: Ticagrelor 90 mg tablet crushed — Ticagrelor 90 mg crushed and suspended in water
  Arms: B
Drug: Dispersed ticagrelor 90 mg tablet suspended in water - nasogastric tube — Dispersed 90 mg ticagrelor 90 mg tablet suspended in water and administered through a nasogastric tube into the stomach
  Arms: C

SUMMARY:
Study to investigate if the uptake of Ticagrelor into the body differs depending on method of administration.

DETAILED DESCRIPTION:
Study to evaluate the bioavailability of the crushed ticagrelor tablets when administered orally or through nasogastric tubes compared to whole ticagrelor tablets given orally

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers aged 18 to 50 years (inclusive) with suitable veins for cannulation or repeated venepuncture
* Have a body mass index between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg (110 pounds [lbs]) and no more than 100 kg (220 lbs).
* Provision of signed and dated, written informed consent prior to any study specific procedures

Exclusion Criteria:

* History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the volunteer at risk because of participation in the study, or influence the results or the volunteer's ability to participate in the study
* History of haemophilia, von Willebrand's disease, lupus anticoagulant or other diseases/syndromes that can either alter or increase the propensity for bleeding
* A personal history of vascular abnormalities including aneurysms; a personal history of severe haemorrhage, haematemesis, melena, haemoptysis, severe epistaxis, severe thrombocytopenia, intracranial haemorrhage; or rectal bleeding within 3 months prior to the screeening visit; or history suggestive of peptic ulcer disease
* History of frequent and/or significant nose bleed or clinically significant non traumatic bleed, bruise/haematoma or any other clinically significant bleeding risk, as judged by the Investigator

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Description of the pharmacokinetic(PK) profile in terms of plasma concentration-time curve (AUC) of ticagrelor | PK samples will be collected pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose
Description of the pharmacokinetic(PK) profile in terms of AUC of the active metabolite of ticagrelor | PK samples will be collected pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose
Description of the pharmacokinetic(PK) profile in terms of maximum plasma concentration (Cmax) of ticagrelor | PK samples will be collected pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose
Description of the pharmacokinetic(PK) profile in terms of Cmax of the active metabolite of ticagrelor | PK samples will be collected pre-dose, 0.5, 1, 2, 3, 4, 6, 8, 10, 12, 16, 24, 36 and 48 hours post-dose

SECONDARY OUTCOMES:
Description of the safety profile in terms of adverse events (AE) | From first dose through to the follow-up visit.
Description of the safety profile in terms of laboratory variables | Safety labs at screening, Day -1, Day 3 (48 hours after treatment) and follow-up
Description of the safety profile in terms of vital signs | Vital signs at screening, pre-dose, 1 h, 3, 6, 12 and 24 hours post-dose, Day 3 for all treatment periods and follow-up
Description of the safety profile in terms of physical examination findings | Physical examination at screening, pre-dose, Day 3 and follow-up
Description of the safety profile in terms of Electrocardiogram (ECG) | ECGs at screening, Day 3 and follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Judith Hsia, MD, Study Director — AstraZeneca, Wilmington, US; Mirjana Kujacic, MD, Study Chair — AstraZeneca Mölndal, Sweden; Saeed Kahn, MBBS, Principal Investigator — Quintiles London, United Kingdom
Locations (1):
- Research Site, London, United Kingdom